CLINICAL TRIAL: NCT02207751
Title: Improving Outcomes in Peritoneal Dialysis: Identification and Characterization of Optimal Clinical Practice to Enhance Peritoneal Dialysis Catheter Functionality, Minimize Access-related Complications and Promote Peritoneal Dialysis as an Initiating Therapeutic Modality for Chronic Kidney Disease.
Brief Title: Improving Outcomes in Peritoneal Dialysis
Status: Withdrawn | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: STH18109
Record Dates: First submitted 2014-07-29; First posted 2014-08-04 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Kidney Disease; Peritoneal Dialysis Access
Keywords: Chronic Kidney Disease; Peritoneal Dialysis Access; Peritoneal Dialysis Catheter; Catheter Function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective is to understand the best way to place Peritoneal Dialysis (PD) catheters, and the best way to collect data regarding their function in England, Wales and Northern Ireland.

Phase 1: We will carry out a detailed examination of existing returned pilot data with emphasis on data fields with poor data completeness and perform root cause analysis, and assess deficiencies in data field definition to identify improvements to be implemented. We will construct and disseminate electronic survey material to all study centres with targeted visits by the Principle Investigator undertaken. These visits will facilitate insight into local organization of data collection including interaction with designated individuals responsible for data returns. PD training days will be organized with emphasis on clinical practice feedback utilizing data acquired in the initial phases. Hospital Episode Statistics will be linked to existing acquired PD patient information to ensure the accuracy of collected data. An online data acquisition system will be developed to allow direct data entry from centres.

Phase 2: On-going and sustained data acquisition performed on a prospective basis.

Phase 3: Primary data analysis including clinical practice variation in England, Wales and Northern Ireland to identify site specific PD catheter functionality variation. Additionally, patient and site specific characteristics that predict clinical outcomes in PD will be identified and characterised.

Phase 4: Clinical guidelines will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (16 years or over) patient requiring first PD catheter placement

Exclusion Criteria:

* Patient less than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All incident patients requiring peritoneal dialysis for end stage renal disease of all etiologies.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Peritoneal dialysis catheter "survival" (sustained function) at 365 days post-insertion (insertion date) | 1 Year
  1. Functional (mechanical) catheter failure
  2. Complication induced catheter failure - Infection, Hemorrhage, Dialysate Leakage & Bowel Perforation

SECONDARY OUTCOMES:
Time to catheter failure | Within 1 Year
  * Catheter failure time (days elapsed from insertion to failure <365 days)
  * Catheter failure time (days elapsed from insertion to failure >365 days)
Missing Data | Baseline & 1 Year
  Missing mandatory data fields
Mortality (all cause) | Within 1 Year
Co-morbid Hospitalization Events | Within 1 Year
  Non-fatal medical events requiring hospitalization, excluding PD related hospitalization
Infection events not resulting in catheter failure | Within 1 Year
  * Exit site / tunnel infection (early): suspected or definite infection around catheter exit site requiring intervention up to 2 weeks following catheter insertion
  * Exit site / tunnel infection (late): suspected or definite infection around catheter exit site requiring intervention after 2 weeks following catheter insertion
  * Peritonitis (early): peritonitis within 2 weeks of catheter insertion
  * Peritonitis (late): peritonitis after 2 weeks following catheter insertion
Leak events not resulting in catheter failure | Within 1 Year
  * Catheter leak events (early): suspected or definite catheter site leak requiring intervention up to 2 weeks following catheter insertion
  * Catheter leak events (late): suspected or definite catheter site leak requiring intervention after 2 weeks following catheter insertion
Modality change | Within 1 Year
  Change of modality from PD to any other form of renal replacement therapy
Catheter non-usage | Within 1 Year
  Catheters inserted but not used for reasons other than failed initial therapy (e.g. Moncrieff)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria R Briggs, MBBS BMedSci, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust